CLINICAL TRIAL: NCT07334249
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Dose-escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of SP-101 Injection Following Single and Multiple Intravenous Doses in Healthy Adult Subjects
Brief Title: First-In-Human (FIH), Single Ascending Dose (SAD) Study and Multiple Ascending Dose (MAD) Study of SP-101 Injection
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Synphatec (Shanghai) Biopharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP-CN_101
Record Dates: First submitted 2025-12-16; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder, Healthy Volunteer
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational Drug group, SP-101 injection (Experimental): Participants will be randomly assigned to the experimental group and placebo groups at ratio of 3:1. Participants assigned to the experimental group will be administered SP-101 by intravenous infusion. Accordingly, participants assigned to the placebo group will be administered placebo by intravenous infusion.
  Interventions: Drug: SP-101 injection
- Placebo group (Placebo Comparator): Participants will be randomly assigned to the experimental group and placebo groups at ratio of 3:1. Participants assigned to the experimental group will be administered SP-101 by intravenous infusion. Accordingly, participants assigned to the placebo group will be administered placebo by intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SP-101 injection — SP-101 is non-competitive antagonist against NMDA receptor and is administered by intravenous infusion.
  Arms: Investigational Drug group, SP-101 injection
Drug: Placebo — Participants will be randomly assigned to the experimental group and placebo groups at ratio of 3:1. Participants assigned to the experimental group will be administered SP-101 by intravenous infusion. Accordingly, participants assigned to the placebo group will be administered placebo by intravenous infusion.
  Arms: Placebo group

SUMMARY:
The goal of this First-In-Human (FIH) trial is to learn about safety, tolerability and pharmacokinetics of single and multiple ascending doses of SP-101 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign written informed consent;
* Aged 18 to 45 years old (inclusive), healthy males or females (male-to-female ratio is 1:1);
* Efficient contraceptive mean required by the protocol, and no plans for fertility, sperm donation or egg donation until 3 months after the last intravenous infusion;
* Body weight:≥50 kg (Male),≥45 kg (Female), Body Mass Index (BMI) of 18 to 28 kg/m2;
* Normal laboratory tests results, physical examination, medical history and surgical history review, 12-lead Electrocardiogram recording, and with no evidence of active and chronic diseases;
* willing and able to comply with all study procedures, restrictions, and visit schedules and to communicate effectively with the investigator;

Exclusion Criteria:

* Individuals with special dietary requirements who cannot adhere to a unified diet (e.g., intolerance to standard meal foods, or those with dysphagia);
* History of intolerance to IV infusion (e.g., severe pain) or unsuitable venous access (e.g., sclerotic, atrophic veins), difficulties with or contraindications to blood sampling; or a history of needle- or blood-injury-related phobia or syncope;
* Lactation or a positive pregnancy test at screening or baseline;
* Any febrile illness or active infection within 14 days prior to the first dose;
* Evidence of drug / substance abuse within the past 5 years, and/or habitual use of any drugs/substances, or a positive urine drug test at screening or baseline;
* Abnormal renal function (eGFR < 90 mL/min/1.73 m²);
* History of QTc prolongation or demonstration of a clinically relevant ECG abnormality at screening;
* Excessive consumption of nicotine products within 3 months prior to screening (average daily cigarette consumption >5 cigarettes), or inability to stop using any tobacco products during the trial, or a positive nicotine test;
* Previous participation in this study; treatment with an investigational product within 30 days prior to study initiation; or planning participation in another clinical trial during the study period;
* Positive test result at screening for any of the following: hepatitis B surface antigen (HBsAg), antibody to hepatitis C virus (anti-HCV), antibody to human immunodeficiency virus (anti-HIV), or treponemal antibody for syphilis;
* Any abnormal results during screening that is deemed clinically significant by the investigator, e.g., resting pulse <55 or >100 bpm; SBP ≥140 or <90 mmHg; DBP ≥100 or <60 mmHg, or ECG, or abnormal laboratory tests results, clinically relevant;
* Significant blood loss (≥200 mL) within 60 days prior to dosing（including trauma, blood sampling, blood donation, etc.）; or planning blood donation during the study or within 30 days post-dose;
* History of alcohol abuse, or average weekly alcohol consumption greater than 14 units within 3 months prior to screening or a positive alcohol breath test at baseline or inability to abstain from alcohol for the duration of the study;
* Excessive daily consumption of tea, coffee, and/or caffeine-rich beverages for a prolonged period within 3 months prior to screening; or intake of xanthine/caffeine-containing or grapefruit-containing foods or beverages (e.g., coffee, strong tea, chocolate, grapefruit) within 24 hours prior to the first intravenous infusion;
* Using any prescription drugs, OTC medications (excluding hormonal contraceptives, topically applied eye/nose drops and creams with no systemic exposure risk), Chinese herbal medicines, or food supplements such as vitamins and calcium supplements within 14 days prior to screening or during the screening period, unless prior approval has been obtained from the Investigator and Sponsor;
* Using any drugs that inhibit or induce the activity of hepatic drug-metabolizing enzymes within 30 days prior to screening;
* History of a major surgical procedure within the past 6 months prior to screening, or planned elective surgery during the course of the study;
* Current or past history of psychiatric and/or , neurological diseases, and abnormalities of the motor or sensory systems, whether confirmed or suspected;
* Any clinically significant disease, or any clinically significant illness, condition, or other finding that, in the investigator's opinion, would pose a risk to subject safety or interfere with the conduct, progress, or completion of the study.;
* History or current using of hallucinations, which is viewed unsuitable for by investigator;
* History or current presence of psychiatric disorders and/or brain dysfunction;
* History of known or suspected hypersensitivity or allergic reaction to any component of the investigational product or to related compounds, drugs, or foods;
* Any other condition or reason that, in the opinion of the Investigator, would make the subject unsuitable for participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-23 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events, throughout study completion | Through study completion, an average of 10 days for SAD and an average of 28 days for MAD

SECONDARY OUTCOMES:
Pharmacokinetic Parameter-AUC₀-inf | From 0 hour before dosing to 72 hours after dosing
  Area under the plasma concentration versus time curve (AUC) from time 0 to infinity
Pharmacokinetic Parameter-AUC₀-last | From 0 hour before dosing to 72 hours after dosing
  Area under the plasma concentration versus time curve (AUC) from time 0 to the last measurable concentration
Pharmacokinetic Parameter-Cmax | From 0 hour before dosing to 72 hours after dosing
  Peak Plasma Concentration (Cmax)
Pharmacokinetic Parameter-Tmax | From 0 hour before dosing to 72 hours after dosing
  Time to reach the Peak Plasma Concentration (Tmax)
Pharmacokinetic Parameter-T½ | From 0 hour before dosing to 72 hours after dosing
  Elimination half life (T½)
Pharmacokinetic Parameter-CL | From 0 hour before dosing to 72 hours after dosing
  Apparent clearance (CL)
Pharmacokinetic Parameter- Vz | From 0 hour before dosing to 72 hours after dosing
  apparent volume of distribution ( Vz)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center (SMHC), Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: WHO website has shared some Background information — https://www.who.int/health-topics/depression#tab=tab_1
- See also: Data and information of the marketed drug (Spravato), the same targeting at NMDAR, have been key reference for study design of this protocol. — https://www.accessdata.fda.gov/drugsatfda_docs/label/2025/211243s019lbl.pdf